CLINICAL TRIAL: NCT06194851
Title: A Randomized Clinical Trial Examining Intranasal Oxytocin Augmentation of Brief Couples Therapy for Veterans With PTSD
Brief Title: Examining Intranasal Oxytocin Augmentation of Brief Couples Therapy for Veterans With PTSD
Acronym: CBCT-OT RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4776-R
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Post-Traumatic Stress Disorder (PTSD)
Keywords: Post Traumatic Stress Disorder (PTSD); Oxytocin; Relational Problems; Brief Cognitive Behavioral Conjoint Therapy; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Eligible dyads will be randomized in a stratified 1:1 manner to the oxytocin or placebo condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, quadruple masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brief Cognitive Behavioral Conjoint Therapy for PTSD plus Intranasal Oxytocin (Experimental): Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) weekly. Prior to each session, the veteran participant will self-administer intranasal oxytocin.
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Brief Cognitive-Behavioral Conjoint Therapy
- Brief Cognitive Behavioral Conjoint Therapy for PTSD plus Intranasal Placebo (Placebo Comparator): Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) weekly. Prior to each session, the veteran participant will self-administer intranasal placebo solution.
  Interventions: Drug: Saline nasal spray; Behavioral: Brief Cognitive-Behavioral Conjoint Therapy

INTERVENTIONS:
Drug: Oxytocin nasal spray — Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each bCBCT session.
  Other Names: Pitocin
  Arms: Brief Cognitive Behavioral Conjoint Therapy for PTSD plus Intranasal Oxytocin
Drug: Saline nasal spray — Veteran participants will self-administer 40 IU of the placebo (intranasal saline spray) 30 minutes before the start of each bCBCT session.
  Arms: Brief Cognitive Behavioral Conjoint Therapy for PTSD plus Intranasal Placebo
Behavioral: Brief Cognitive-Behavioral Conjoint Therapy — Eight sessions of standardized bCBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
  Other Names: bCBCT

SUMMARY:
Leveraging veterans' intimate relationships during treatment for posttraumatic stress disorder (PTSD) has the potential to concurrently improve PTSD symptoms and relationship quality. Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) is a manualized treatment designed to simultaneously improve PTSD and relationship functioning for couples in which one partner has PTSD. Although efficacious in improving PTSD, the effects of CBCT on relationship satisfaction are small, especially among Veterans. Pharmacological augmentation of bCBCT with intranasal oxytocin, a neurohormone that influences mechanisms of trauma recovery and social behavior, may help improve the efficacy of bCBCT. The purpose of this randomized placebo-controlled trial is to compare the clinical and functional outcomes of bCBCT augmented with intranasal oxytocin (bCBCT + OT) versus bCBCT plus placebo (bCBCT + PL). The investigators will also explore potential mechanisms of action: communication, empathy, and trust.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the effects of Brief Cognitive Behavioral Conjoint Therapy (bCBCT) paired with intranasal oxytocin (OT) versus placebo on PTSD symptoms, intimate relationship satisfaction and psychosocial functioning in a sample of veterans with PTSD (across all measures) and their intimate partners (relationship satisfaction only). The study will also explore the impact of intranasal oxytocin on potential mechanisms of action (i.e., communication skills, empathy, and trust).

bCBCT is a modified PTSD-specific cognitive-behavioral psychotherapy attended by the couple that uses close relationships as the vehicle for recovery. Across eight 75-minute sessions, this manualized therapy addresses the patient's PTSD and relationship functioning simultaneously via its focus on PTSD psychoeducation within relationship contexts, communication skills, behavioral approach exercises, and cognitive interventions.

Oxytocin is a 9-amino-acid nonapeptide hormone produced by the paraventricular and supraoptic nuclei of the hypothalamus that regulates human emotions, social cognition, and social behaviors. Oxytocin is released to several brain areas, including the amygdala, hypothalamus, hippocampus, insula, and striatum, and effects are mediated by oxytocin receptors found in these regions.

Intranasal administration of oxytocin may offer understanding of the causal effects of oxytocin on human behavior. Intranasal oxytocin is safe and easy to administer, with a short half-life that makes it highly suitable for adding to behavioral interventions. Intranasal oxytocin is best known for its widespread effects on affiliative processes and behaviors. For example, intranasal oxytocin increases trust, empathy, generosity, positive communication, and emotional disclosure. Oxytocin also improves social cognition, including emotion recognition and empathic accuracy. The combination of intranasal oxytocin with provision of social support suppresses cortisol release and subjective responses to social stress.

Intranasal oxytocin can be conceptualized as a "psychotherapy process catalyst", in that oxytocin could enhance patients' openness to intervention, attention to others' communication, and willingness and ability to develop therapeutic alliance. A recent systematic review of 14 studies of the effects of intranasal oxytocin on PTSD symptoms concluded that there is tentative evidence for the clinical utility of intranasal oxytocin for PTSD, although more studies with chronic administration among clinical samples are needed.

The investigators will employ a double blind, placebo-controlled RCT design in which Veterans will receive a dose of oxytocin or placebo before each bCBCT session and complete mid-treatment, post-treatment, 3-month, and 6-month follow-up assessments. Based on the findings from past bCBCT trial and the investigators' recent bCBCT + OT pilot study, the investigators anticipate about 1/3 of the sample will be dual Veterans or the identified Veteran is female. The investigators project an approximate 20-25% attrition rate, resulting in approximately 100 couples completing treatment. Consistent with past trials, to enhance retention, the investigators will ask couples to provide contact information for collateral informants who can reach them if the investigators are unable to do so via their primary contact information. Study personnel will routinely remind couples of appointments via telephone and/or letters and the team will meet weekly to review and problem-solve retention strategies. These are all established procedures implemented from successful prior trials. If successful, the study will advance knowledge of strategies for improving Veterans' quality of life by improving their intimate relationships along with PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Veteran:

1. Be a Veteran (age 18 or older) with a current DSM-5 diagnosis of PTSD (as assessed by the CAPS-5 with a minimum severity score of 25) no less than 3 months after the index trauma occurred (to allow for potential natural recovery)
2. Be on a stable psychoactive medication regimen for at least 4 weeks (if applicable)
3. Be enrolled and eligible to receive care at the VASDHS

   Inclusion criteria for Partner:
4. Be an intimate partner (age 18 or older) who is willing to participate in the intervention (partners can also be Veterans but cannot meet criteria for possible PTSD per the PCL-5)

   Inclusion criteria for Veteran and Partner:
5. Be married, or cohabitating for at least 6 months
6. Willing to be randomized into either treatment condition (bCBCT + OT or bCBCT + PL)
7. Agree to have assessment and treatment sessions audio/video recorded
8. Agree not to receive other individual trauma-focused psychotherapy for PTSD or any form of conjoint therapy during the treatment portion of the study
9. Have the capacity to participate in virtual care (access to internet via DSL or a cable provider, private space)

   Exclusion Criteria:

   Exclusion criteria for Veteran and Partner:
10. Current substance dependence in either member of the couple not in remission for at least 3 months, as assessed by the Alcohol Use Disorders Identification Test (AUDIT)74 and Drug Abuse Screening Test (DAST)75
11. Any current uncontrolled psychotic disorder in either member of the couple as assessed by positive screen on the Prime Screen-Revised (PS-R). Exclusion to be determined following case consult by PI or other clinician.
12. Imminent suicidality or homicidality in either member of the couple (e.g., C-SSRS)
13. Any severe cognitive or medical impairment in either member of the couple making it difficult to regularly attend weekly couples psychotherapy
14. Any perpetration of severe physical or sexual relationship aggression (as assessed by the CTS-2) or fear/intimidation (3-item IPV screen, Couples Questionnaire) in the past year

    Exclusion criteria for Veteran:
15. Severe ongoing medical problems, including heart disease, uncontrolled hypotension (systolic blood pressure <100 mm Hg) or hypertension (systolic BP >130 or diastolic BP > 80 mm Hg), and neuroendocrinological disorders (e.g., diabetes). Exclusion to be determined in collaboration with study physician following completion of physician's one-on-one appointment with Veteran and review of all relevant information (e.g., risk factors, health history, concomitant medications, etc.) from Veteran's VA medical record and study screening/assessment processes including selfreport measures and blood pressure measurement. Additionally, Veterans for whom the study physician has elevated concern, will be asked to attend an in-person visit at a VA medical center, clinic, or the Veterans Medical Research Foundation before enrollment.
16. Positive screen (7+) for borderline personality disorder (BPD) as assessed by the MacLean Screening Instrument for BPD76. Exclusion to be determined following case consult by PI or other clinician.
17. Pregnancy, delivery in the past 6 months, current breastfeeding, or the ability to become pregnant while not practicing an effective method of contraception. If able to become pregnant, Veteran must have a highly sensitive negative urine pregnancy test verified visually via telehealth or in-person at the Veterans Medical Research Foundation by research staff at study entry and prior to each medication administration during treatment. Veteran must verbally confirm that they completed the test themselves that day. Veteran must also agree to use an effective birth control method from study entry until conclusion of treatment to prevent pregnancy. The ability to become pregnant is defined as: assigned female at birth, fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

    Effective birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, oral hormones, a barrier contraception method (e.g., male or female condoms, diaphragm, cap), or vasectomized sole sexual partner.

    Pregnancy tests will be purchased by the study and mailed to Veteran unless PI has approved waiver of testing requirement.
18. Known allergy to preservatives (i.e., Methylparaben, Propylparaben, Glycerin, Sodium Benzoate, Potassium Sorbate, and Disodium EDTA) utilized in oxytocin nasal spray.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
PTSD diagnosis and severity change | Baseline - 6-months post treatment
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 20-item diagnostic interview administered by trained evaluators to assess PTSD in a participant. Based on DSM-5 diagnostic criteria, evaluators ask about the severity of four PTSD-related symptom clusters: re-experiencing, avoidance, negative alterations in cognition and mood, and alterations in arousal and reactivity. The evaluator rates responses on a 5-point Likert scale (0 = Absent to 4 = Extreme/Incapacitating). Total scores range from 0 to 80 with higher scores indicating greater severity. CAPS-5 will be completed by veterans with PTSD only.

SECONDARY OUTCOMES:
Relationship satisfaction | Baseline - 6-months post treatment
  The Couples Satisfaction Index (CSI-32). The CSI-32 is a 32-item self-report survey that measures romantic relationship satisfaction. The first item measures the overall happiness of the relationship on a 7-point scale (0 = Extremely unhappy to 6 = Perfect). The other 31 items capture satisfaction, quality, and happiness of the relationship on 6-point scales (0 to 5) with varying response options. Total CSI-32 scores range from 0 to 161 with higher scores indicating greater relationship satisfaction. Scores below 104.5 indicate clinical relationship distress. CSI-32 will be completed by both partners.

OTHER OUTCOMES:
Psychosocial functioning | Baseline - 6-months post treatment
  The Brief Inventory of Psychosocial Functioning (B-IPF) is a brief version of the Inventory of Psychosocial Functioning (IPF) that measures functioning impairment across seven domains: intimate relationships, family and parenting, friendships, work, socializing, education, and self-care over the past 30 days. Total scores, ranging from 0 to 100, are calculated as the sum score divided by the total possible score multiplied by 100, with higher scores indicating greater impairment in functioning. B-IPF will be completed by veterans with PTSD only.
Trust | Baseline - 6-months post treatment
  The Trust in Close Relationships Scale (TCRS) is a 17-item self-report measure of trust in close relationships, including predictability, dependability, and faith in close others. The TCRS uses a 7-point Likert scale (-3 = Strongly Disagree to 3 = Strongly Agree) to capture one's level of trust in their intimate partner. Total TCRS scores range from -51 to 51, with higher scores indicating higher levels of trust. The TCRS will be completed by both partners.
Empathy | Baseline - 6-months post treatment
  The Interpersonal Reactivity Index for Couples (IRIC) is a measure of empathy expressed within romantic relationships. The IRIC is a 28-item self-report assessment in which participants select their responses to each item on a 5-point Likert scale (0 = does not describe me well to 4 = describes very well). Items are divided into four subscales with 7 items each: perspective-taking, fantasy, empathic concern, and personal distress. Total scores on the IRIC range from 0 to 112 with higher scores indicating higher empathy. This measure will be completed by both partners.
Communication | Baseline - 6-months post treatment
  The Brief Communication Skills Test (CST) is a self-report measure of communication skills that was created by pulling the positive communication questions from the full CST. Participants rate items on a 7-point scale from 1 (Almost Never) to 7 (Almost Always). Total scores range from 10 to 70, with higher scores indicating more positive communication. This will be completed by both partners.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A. Morland, PsyD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA; Lauren M. Sippel, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sippel LM, Wachsman TR, Kelley ME, Knopp KC, Khalifian CE, Maglione JE, Glynn SM, Macdonald A, Monson CM, Flanagan JC, Holtzheimer PE, Morland LA. Design of a randomized clinical trial of brief couple therapy for PTSD augmented with intranasal oxytocin. Contemp Clin Trials. 2024 Jun;141:107534. doi: 10.1016/j.cct.2024.107534. Epub 2024 Apr 12. PMID 38614447